CLINICAL TRIAL: NCT05088525
Title: Meniscal Root Tears: Evaluating Meniscal Extrusion After Root Repair with and Without Transtibial Peripheral Stabilization Sutures Using Ultrahigh Magnetic Fields: a Randomized Controlled Trial
Brief Title: Meniscal Root Tears: Evaluation Using an Ultrahigh MRI
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Twin Cities Orthopedics (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: RFL_UMN-7T MRI
Record Dates: First submitted 2021-09-14; First posted 2021-10-22 (Actual); Last update posted 2024-11-22 (Actual); Status verified 2024-11

CONDITIONS: Knee Injuries
Keywords: Meniscal Root; MRI
MeSH Terms: conditions — Knee Injuries

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Two-tunnel meniscal root repair without a peripheral stabilization suture (Active Comparator): Standard root repair surgery.
  Interventions: Procedure: MRI
- Meniscal root repair with an additional transtibial peripheral stabilization suture (Experimental): Meniscus root repair with an added stabilization suture
  Interventions: Procedure: MRI

INTERVENTIONS:
Procedure: MRI — MRI for standard of care meniscus root repair surgery - noting with an added stabilization suture if it is able to successfully slow down the progression of osteoarthritis versus a standard root repair surgery.

SUMMARY:
Meniscal root tears have been recently recognized to be one of the most common causes for the progression of arthritis in relatively young patients. The purpose of the study will be to assess if the addition of a transtibial peripheral stabilization suture helps to decrease both meniscal extrusion and if it helps to decrease the progression of osteoarthritis of the medial compartment of the knee in the early timeframe postoperatively.

DETAILED DESCRIPTION:
Studies have reported that the most common reason why patients require total knee arthroplasty before the age of 60 is a neglected or meniscectomized medial meniscus root tear. Overall, it has been noted that meniscal root repairs are cost effective and that the outcomes of meniscus root repairs are demonstrating patients have a significant improvement of their preoperative symptoms up to several years after surgery. Because most centers have only been preforming meniscus root repairs over the last five to ten years, we are now starting to recognize why some of the repairs do not function as well as others. The number one reason appears to be due to a postoperative meniscus extrusion. Meniscus extrusion has been seen in up to 50% of postoperative patients, and biomechanical studies have demonstrated that the cushioning effect of the medial meniscus does not function as well when there is a meniscus extrusion present. New biomechanical studies have demonstrated that the addition of a peripheral stabilization suture at the far posteromedial aspect of the medial tibial plateau helps to hold the meniscus better in the joint and that it also results in a significant decrease in load on the medial compartment. However, clinical studies are lacking to date as to whether a peripheral stabilization suture may or may not improve the protected function of the medial meniscus, decreased extrusion, and potentially lead to a less amount of progression of osteoarthritis in the medial compartment of the knee.

Therefore, this study strives to both assess the ability of a meniscus root repair to slow down the progression of arthritis of the medial compartment of patients with a 7-Tesla MRI scanner and also to concurrently assess the ability of the usage of a transtibial peripheral stabilization suture to decrease or eliminate meniscal extrusion. The importance of this study is that if the peripheral stabilization suture is noted to both decrease the progression of arthritis and also to decrease the meniscus extrusion, it will be a significant step forward in the treatment of these complex meniscal tears.

ELIGIBILITY:
Inclusion Criteria:

* Between ages 14-70 years old
* Has suspected meniscus root tear
* Able to consent for themselves for adults
* English speaking
* Males or females
* Is willing and able to comply with the clinical trial plan and able to understand and sign the Patient Informed Consent Form.

Exclusion Criteria:

* < 14 years old or open physes
* >70 years old
* Pregnant
* Previous or concurrent vascular injury (vascular bypass procedure)
* Associated fractures requiring concurrent surgery
* Found to have contraindications to MRI based on a systematic safety screening developed by the CMRR

Ages: 14 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 27 (Actual)
Dates: Start 2020-11-20 (Actual); Primary Completion 2024-11-15 (Actual); Study Completion 2024-11-15 (Actual)

PRIMARY OUTCOMES:
MRI | Pre-operatively
  Musculoskeletal radiologist assessment of medial meniscus extrusion and cartilage specific sequences gathered
MRI | 6 months post-operatively
  Musculoskeletal radiologist assessment of medial meniscus extrusion and cartilage specific sequences gathered

SECONDARY OUTCOMES:
visual analog scale (VAS) scores | pre-operatively and post-operatively at 3 and 6 months
  Pain scale 0-100
International Knee Documentation Committee (IKDC) | pre-operatively and post-operatively at 3 and 6 months
  The questionnaire looks at 3 categories: symptoms, sports activity, and knee function. Scores are obtained by summing the individual items, then transforming the crude total to a scaled number that ranges from 0 to 100. The higher the score, better outcomes 87/87 = 100%
Cincinnati Knee Rating System | pre-operatively and post-operatively at 3 and 6 months
  Functional assessment based on 6 abilities important for participation in sports. The higher the score, better outcomes 100/100 = 100%
Knee injury and Osteoarthritis Outcome Score (KOOS) | pre-operatively and post-operatively at 3 and 6 months
  Assesses five outcomes: pain, symptoms, activities of daily living, sport and recreation function, and knee-related quality of life. The maximum score a patient can achieve is 100, indicating no knee problems.
Tegner | pre-operatively and post-operatively at 3 and 6 months
  the higher the score, better outcomes 100/100 = 100% The scale is numbered on a "0-10" format, with 1 being professional and 1 being a person who is disabled from knee issues.
Lysholm Knee Scoring Scale | pre-operatively and post-operatively at 3 and 6 months
  Consists of eight items that measure: pain (25 points), instability (25 points), locking (15 points), swelling (10 points), limp (5 points), stair climbing (10 points), squatting (5 points), and need for support (5 points). Every question response has been assigned an arbitrary score on an increasing scale. The total score is the sum of each response to the eight questions, and may range from 0-100.
Veterans Rand 12 (VR-12) General Health Survey | pre-operatively and post-operatively at 3 and 6 months
  VR-12 includes 12 original question items from the VR-36. The questions in this survey correspond to seven different health domains: general health perceptions, physical functioning, role limitations due to physical and emotional problems, bodily pain, energy/fatigue levels, social functioning and mental health. Answers are summarized into two scores, a Physical Component Score (PCS) and a Mental Component Score (MCS) which then provides an important contrast between the respondents' physical and psychological health status. The higher the score, better outcomes
Lower extremity functional scale | pre-operatively and post-operatively at 3 and 6 months
  Questionnaire containing 20 questions about a person's ability to perform everyday tasks. The LEFS can be used by clinicians as a measure of patients' initial function, ongoing progress and outcome, as well as to set functional goals. The columns on the scale are summed to get a total score. The maximum score is 80. The higher the score, better outcomes = 80/80 =100%
Sports Medicine Questionnaire | pre-operatively and post-operatively at 3 and 6 months
  Assess return to activity; no scale, individual questions
Patient satisfaction | Post-operatively at 3 and 6 months
  0- 100, higher the score, the better

CONTACTS AND LOCATIONS:
Overall Officials: Robert F LaPrade, MD, PhD, Principal Investigator — Twin Cities Orthopedics
Locations (1):
- Twin Cities Orthopedics, Edina, Minnesota, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Tollefson LV, Kajabi AW, Hedayati E, Knutsen K, Takahashi T, Ellermann J, LaPrade RF. Medial Meniscal Extrusion Increased on 6-Month Magnetic Resonance Imaging, Despite Successful Posterior Root Repair With or Without a Centralization Suture: A Randomized Controlled Clinical Trial. Am J Sports Med. 2025 Oct;53(12):2808-2816. doi: 10.1177/03635465251366443. Epub 2025 Sep 3. PMID 40901697